CLINICAL TRIAL: NCT02017275
Title: A Prospective, Multicenter, RAndomized, CoNtrolled, Study Comparing the Safety and Efficacy Between BuMA eG Based BioDegradable Polymer Stent and EXCEL Biodegradable Polymer Sirolimus-eluting Stent in "ReAl-World" Practice (PANDA-III)
Brief Title: Comparison of BuMA eG Based BioDegradable Polymer Stent With EXCEL Biodegradable Polymer Sirolimus-eluting Stent in "Real-World" Practice
Acronym: PANDA-III
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sino Medical Sciences Technology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PANDA-Ⅲ
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BuMA group (Experimental): Implant BuMA stent only
  Interventions: Device: BuMA
- EXCEL group (Active Comparator): Implant EXCEL stent
  Interventions: Device: EXCEL

INTERVENTIONS:
Device: BuMA — This group will contain 1175 subjects.
  Arms: BuMA group
Device: EXCEL — This group will contain 1175 subjects.
  Arms: EXCEL group

SUMMARY:
PANDA III is sought to investigate the safety and efficacy of a PLGA-polymer with electro-grafting base layer sirolimus-eluting stent (SES) versus a PLA-polymer SES at 12 months follow-up.

DETAILED DESCRIPTION:
The BuMA stent (SINOMED, Beijing, China) was a novel biodegradable PLGA polymer sirolimus-eluting stent (SES), with design of adding an electro-grafting (eG) base layer between the polymer and the stainless steel stent strut.The eG layer can secure adhesion of the biodegradable PLGA coating as a result of the interdigitation, and the PLGA coating ensures 100% drug release within 30 days.The initial investigation showed a high strut coverage rate in both the BuMA stent and the Xience V stent at 3 months follow-up. Moreover, earlier vascular healing after drug-eluting stent implantation may reduce the incidence of stent thrombosis at follow-up and potentially shorten dual antiplatelet therapy duration. Therefore, we performed this randomized trial to investigate 12 months target lesion failure between the BuMA and the EXCEL stent, both with same eluted drug sirolimus, however different biodegradable polymer carriers.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 of age;
* Symptomatic ischemic heart disease and/or objective evidence of myocardial ischemia including chronic stable coronary artery disease, or acute coronary syndrome including non-ST-elevation and ST-elevation myocardial infarction;
* Acceptable candidate for CABG;
* The patient is willing to comply with specified follow-up evaluations;
* Patients who agree to accept the follow-up visits.
* Patients can understand the study objectives psychologically and linguistically and show the sufficient compliance to the study protocol. Patients present acceptance of the risks and benefits described in the informed consent form.
* At least one lesion with a diameter stenosis >50% or more suitable for coronary stent implantation in a vessel with a reference diameter ranging from 2.5 mm to 4.0 mm;

Exclusion Criteria:

* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure.
* Patient has other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than 1 year);
* Patient has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, stainless steel alloy, cobalt chromium, rapamycin , styrene-butylenes-styrene or poly-lactic acid (PLA) polymer, and/or contrast sensitivity that cannot be adequately pre-medicated;
* Any significant medical condition which in the Investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in another investigational drug or device study or patient in inclusion in another investigational drug or device study during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2348 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Target lesion failure (a composite of cardiac death, target lesion myocardial infarction and ischemia driven target lesionsrevascularization TLR) at 1 year | 12 months after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, Dr, Principal Investigator — Fuwai Hospital, Chinese Academy of Medical Science
Locations (1):
- Fuwai hospital, Beijing, China

REFERENCES:
- [Derived] He J, Bian X, Zhang R, Yuan S, Guan C, Zou T, Liu L, Song C, Xie L, Wang H, Qiao Z, Yin D, Xu B, Dou K. Impact of Relative Improvement in Quantitative Flow Ratio on Clinical Outcomes After Percutaneous Coronary Intervention - A Subanalysis of the PANDA III Trial. Circ J. 2024 May 24;88(6):921-930. doi: 10.1253/circj.CJ-22-0743. Epub 2024 Jan 27. PMID 38143084
- [Derived] Zhang R, Wu S, Yuan S, Guan C, Zou T, Qiao Z, Xie L, Wang H, Song L, Xu B, Dou K. Effects of diabetes mellitus on post-intervention coronary physiological assessment derived by quantitative flow ratio in patients with coronary artery disease underwent percutaneous coronary intervention. Diabetes Res Clin Pract. 2022 Apr;186:109839. doi: 10.1016/j.diabres.2022.109839. Epub 2022 Mar 21. PMID 35331810
- [Derived] Zhang R, Xu B, Dou K, Guan C, Zhao Y, Wang X, Zou T, Qiao Z, Xie L, Wang H, Yuan S, Song L, Tu S, Wang Y, Wijns W. Post-PCI outcomes predicted by pre-intervention simulation of residual quantitative flow ratio using augmented reality. Int J Cardiol. 2022 Apr 1;352:33-39. doi: 10.1016/j.ijcard.2022.01.054. Epub 2022 Jan 31. PMID 35101540
- [Derived] Zhang R, Dou K, Guan C, Zou T, Zhang M, Yuan S, Qiao Z, Xie L, Sun Z, Song L, Qiao S, Stone GW, Xu B. Outcomes of quantitative flow ratio-based percutaneous coronary intervention in an all-comers study. EuroIntervention. 2022 Feb 18;17(15):1240-1251. doi: 10.4244/EIJ-D-21-00176. PMID 34219669
- [Derived] Zhang R, Song C, Guan C, Liu Q, Wang C, Xie L, Sun Z, Cai M, Zhang M, Wang H, Liu J, Dou K, Xu B. Prognostic Value of Quantitative Flow Ratio Based Functional SYNTAX Score in Patients With Left Main or Multivessel Coronary Artery Disease. Circ Cardiovasc Interv. 2020 Oct;13(10):e009155. doi: 10.1161/CIRCINTERVENTIONS.120.009155. Epub 2020 Oct 12. PMID 33040580
- [Derived] Jia S, Guan C, Yuan J, Cao X, Qin L, Li Y, Li Z, Nie S, Hou S, Zhang M, Brouwer M, Suryapranata H, Xu B, Gao R. Two-year safety evaluation of a biodegradable polymer sirolimus-eluting stent with increased drug elution and polymer absorption kinetics in complex patient and lesion cohort. Catheter Cardiovasc Interv. 2020 Feb;95(2):206-215. doi: 10.1002/ccd.28288. Epub 2019 Apr 16. PMID 30990245
- [Derived] Wang J, Guan CD, Yuan JS, Gao RL, Xu B, Qiao SB. [Prognostic value of SYNTAX score on 1 year outcome in patients underwent percutaneous coronary intervention]. Zhonghua Xin Xue Guan Bing Za Zhi. 2018 Apr 24;46(4):267-273. doi: 10.3760/cma.j.issn.0253-3758.2018.04.004. Chinese. PMID 29747321
- [Derived] Xu B, Gao R, Yang Y, Cao X, Qin L, Li Y, Li Z, Li X, Lin H, Guo Y, Ma Y, Wang J, Nie S, Xu L, Cao E, Guan C, Stone GW; PANDA III Investigators. Biodegradable Polymer-Based Sirolimus-Eluting Stents With Differing Elution and Absorption Kinetics: The PANDA III Trial. J Am Coll Cardiol. 2016 May 17;67(19):2249-2258. doi: 10.1016/j.jacc.2016.03.475. PMID 27173037